CLINICAL TRIAL: NCT01763892
Title: Physiologic Mechanisms in Pediatric Traumatic Brain Injury (TBI)
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00040284; 71244 (Other Grant/Funding Number: RWJF); 1P30NR014139-01 (NIH)
Record Dates: First submitted 2012-11-30; First posted 2013-01-09 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Traumatic Brain Injury
Keywords: Pediatric; Traumatic Brain Injury; TBI; Apolipoprotein E; apo-E; Vasospasm; Genetics; Physiologic Mechanisms; Neurocognitive Outcomes; Endothelin 1
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Apolipoprotein E (apo-E) genotype/SNPs Endothelin 1 genotype/SNPs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children admitted to hospital with a TBI: non-intervention study

SUMMARY:
The aims of this study explore the relationships between cerebral vasospasm, apolipoprotein-E (apo-E) genotype, physiologic symptoms, and neurocognitive outcomes that may either intensify or ameliorate secondary injury, for children with a traumatic brain injury. Exploring the apo-E genotype will help us know if injury response is altered in certain children and will aid in developing interventional approaches.

DETAILED DESCRIPTION:
The purpose of this study is to advance knowledge of neurocognitive outcomes in pediatric traumatic brain injury (TBI) patients by exploring the relationships between physiologic factors of cerebral vasospasm, apolipoprotein E (apo-E) allele, biomarkers, and neurocognitive outcomes. This study is a funded project within Duke University School of Nursing National Institutes of Health/National Institute of Nursing Research (NIH/NINR) P30 Center of Excellence Grant. This study will continue on with some of the work of a small intramural grant study determining the feasibility of conducting pediatric TBI research at DUHS. It will advance the measurement of vasospasm by translating the use of the Transcranial Doppler (TCD) ultrasound to neuromonitoring in children. To date, this will be the first pediatric study examining the relationship of cerebral vasospasm, apo-E, and biomarkers with neurocognitive outcomes. Unlike adult TBI patients, cerebral vasospasm, apo-E, and biomarker collections have yet to be examined in pediatric neurotrauma patients in the Duke University Health System. Although neurocognitive outcomes are a standard of care for TBI patients at Duke University Health System (DUHS), the data has yet to be examined within the realm of pediatric neurodiagnostic physiologic measures. By obtaining preliminary data in 35 patients, it will allow for the evaluation of multi-diagnostic measures in pediatric TBI patients, as well as provide data for future funding for a larger regionally-scale study.

ELIGIBILITY:
Inclusion Criteria:

1. TBI patients admitted to the pediatric intensive care service (PICU)or pediatric progressive care unit
2. Range in age from birth to 15 years
3. TBI with a Glasgow Coma Scale of 3-15
4. Acoustic window for adequate transcranial doppler (TCD) ultrasound
5. English or Spanish speaking or understanding parent/legal guardian to consent
6. Access for a buccal swab for genotyping

Exclusion Criteria:

1. Non-English or Spanish speaking parents/legal guardian
2. Children with a previously diagnosed neurodevelopmental delay

Ages: 5 Days to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Presence of apolipoprotein E (apo-E) allele | Day 1
  Collection of Apo-E allele will be obtained by buccal swab upon enrollment

SECONDARY OUTCOMES:
Vasospasm detection by Transcranial Doppler Ultrasound (TCD) | 8 days
  Daily Transcranial doppler ultrasound will performed in pediatric traumatic brain injury patients through hospital day 8. If vasospasm is present and persists beyond hospital day 8, daily TCD examinations will be continued until resolution of vasospasm is noted.

OTHER OUTCOMES:
Biomarker Detection | 5 days
  Detection of a defined set of protein biomarkers from biological samples collected at baseline, 24, 48, and 96 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Karin Reuter-Rice, PhD, Principal Investigator — DUSON
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States